CLINICAL TRIAL: NCT06961617
Title: Safety and Efficacy of Autologous HBV-TCR T Cell Therapy (LioCyx-M) for the Treatment of Hepatocellular Carcinoma
Brief Title: Autologous HBV-TCR T Cell Therapy (LioCyx-M) for the Treatment of Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lion TCR Pte. Ltd. (Industry)
Collaborators: Beijing GoBroad Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTCR-HCC-3-6
Record Dates: First submitted 2025-05-06; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LioCyx-M (Experimental): LioCyx-M, HBV antigen-specific TCR-redirected T cells, will be administered every week at a dose of 5-10 x 10^6 cells/kg body weight (BW).
  Interventions: Drug: LioCyx-M, HBV antigen-specific TCR-redirected T cells

INTERVENTIONS:
Drug: LioCyx-M, HBV antigen-specific TCR-redirected T cells — Via intravenous (IV) infusion

SUMMARY:
This is a single center and open-label study to determine the safety and efficacy of mRNA HBV-TCR redirected T-cells in HBV-related HCC who are not amenable to/failed conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosis confirmed by histology/ cytology or clinically
* HCC that is not amenable to curative surgical and/or locoregional therapies, or progressive disease after surgical and /or locoregional therapies
* Has failed at least one line of systemic therapy for HCC
* ECOG performance status ≤1
* Serum HBsAg positivity
* Child-Pugh A (5 - 7 points)
* Life expectancy of at least 1 year
* HLA profile: HLA-A*02:01 or HLA-A*24:02

Exclusion Criteria:

* Brain metastasis
* Second primary malignancy that is clinically detectable at the time of consideration for study enrolment, except for in situ carcinoma of the cervix, non-melanoma skin carcinoma localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer and superficial bladder tumors
* Concurrent administration of any other anti-tumour therapy, including cytotoxic chemotherapy, TKI therapy, and immunotherapy.
* Use of any investigational product (IP) or investigational medical device within 28 days of study drug administration
* Serum HBV DNA levels ≥ 200 IU/ml at screening
* Serum HBsAg levels ≥ 10,000 IU/ml at screening
* Women who are pregnant or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessments of adverse events/serious adverse events | Start of treatment until 28 days post last dose
  To evaluate the safety of LioCyx-M
Objective Response Rate (ORR) | Up to 2 years
  To evaluate the anti-tumor efficacy of LioCyx-M

SECONDARY OUTCOMES:
Duration of Response (DoR) | Up to 2 years
  To evaluate the anti-tumor efficacy of LioCyx-M
Progression Free Survival (PFS) | Up to 2 years
  To evaluate the anti-tumor efficacy of LioCyx-M
Overall Survival (OS) | Up to 2 years
  To evaluate the anti-tumor efficacy of LioCyx-M

CONTACTS AND LOCATIONS:
Overall Officials: Tina Wang, Study Director — Lion TCR Pte. Ltd.
Locations (1):
- Gaobo Boren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No